CLINICAL TRIAL: NCT04836741
Title: Comparision of the Outcomes and Learning Curve of Rectectomy for Rectal Cancer Using Diverse Minimally Technologies: Surgical Robot "Micro Hand S", Laparoscope
Brief Title: Chinese Surgical Robot Clinical Study on Rectectomy for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XY3-DSRCS1507A02
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Laparoscopes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro Hand S robot-assisted surgery (Experimental): This group is consisted of 40 cases performed using the Micro Hand S robot by one single surgeon for rectal cancer
  Interventions: Device: Micro Hand S robot
- Laparoscopic surgery (Active Comparator): This group is consisted of 65 cases performed using the laparoscope by one single surgeon for rectal cancer
  Interventions: Device: Laparoscope

INTERVENTIONS:
Device: Micro Hand S robot — The surgeries are performed with the Micro Hand S robot
  Arms: Micro Hand S robot-assisted surgery
Device: Laparoscope — The surgeries are performed with the laparoscope
  Arms: Laparoscopic surgery

SUMMARY:
Central South University in collaboration with Tianjin University developed the first domestically produced Chinese minimally invasive surgical (MIS) robot system which named "Micro Hand S" in 2013. This new MIS robot had been authorized to enter the clinical trial stage by the Ethics Committee of the Third Xiangya Hospital at Central South University. The Micro Hand S robot is safe and feasible in the preliminary study. However, compared with minimally invasive approaches (da Vici, laparoscope), the merits and demrits of rectectomy for rectal cancer are unclear. Therefore, the investigators conduct this retrospective study to focus on this concern.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed rectal cancer; ASA score < 3

Exclusion Criteria:

* palliative resections, combined resections, distant metastasis, a previous history of abdominal/or pelvic surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Type of surgical procedure | up to 1 week after operation
  It was defined as what type of procedure was pferformed, for example, low anterior, abdominal perineal resection
Operative time (min) | up to 1 week after operation
  It was defined as the duration from skin incision to skin closure
Conversion | up to 1 week after operation
  Conversion was defined as any change in strategy to open surgery
Bloos loss (ml) | up to 1 week after operation
  It was defined as the amount of blood in the whole surgical time
Protective ileostomy | up to 1 month after operation
  It was defined as ileostomy which diverted the feces to To ensure anastomotic healing
Hospital stay (day) | up to 1 month after operation
  It was defined as the length of hospital stay
Tumor size (cm) | up to 1 month after operation
  It was defined as the longitudinal diameter of the tumor
Retrieved lymph node | up to 1 month after operation
  It was defined as the number of all the lymph nodes for each patien
pTNM stage | up to 1 month after operation
  It was defined as the pathological stage of the tumor according the TNM classification
Length of distal ressction margin (cm) | up to 1 month after operation
  It was defined as the distance betwen the distal resection margin and the low margin of the tumor
Status of the surgical margin | up to 1 month after operation
  It was defined as whether the distal and circumferential resection margins was involved the tumor cell under microscope
Quality of specimen | up to 1 month after operation
  The quality of the speciman was graded according to the protocol proposed by Quirke
Postoperative complication | up to 1 month after operation
  It was defined as the adverse events after operation and the complications were classfied according to the Clavien-Dindo (C-D) classification
International Prostate Symptom Score | at least12 months after operation
  It assessed the urination with 7 items
International Index of Erectile Function | at least 12 months after operation
  It assessed erectile function with 5 items
Local recurrence | at least 1 years after operation
  It was defined as the tumor was again found in the pelvic cavity
Disease free survival | at least 1 years after operation
  It was defined as the duration between the operation and date of the tumor recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Wang G, Li Z, Ling H, Yi B, Zhu S. Comparison of the operative outcomes and learning curves between laparoscopic and "Micro Hand S" robot-assisted total mesorectal excision for rectal cancer: a retrospective study. BMC Gastroenterol. 2021 Jun 7;21(1):251. doi: 10.1186/s12876-021-01834-1. PMID 34098897